CLINICAL TRIAL: NCT02818894
Title: Comparison of Lidocaine Versus Bupivacaine Spinal Anesthesia in Total Hip Arthroplasty: A Randomized, Double-Blind, Prospective Study
Brief Title: Spinal Anesthesia in Total Hip Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated due to pressing matters related to the COVID-19 pandemic - staff shortages and changes of personnel, data gaps due to the pandemic, participants not being able to continue follow-up visits, and ongoing enrollment issues.
Sponsor: Thomas L Bradbury (Other)
Responsible Party: Sponsor-Investigator, Thomas L Bradbury, Associate Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00083867
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Results first posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-08

CONDITIONS: Total Hip Arthroplasty
Keywords: Hip replacement; Total hip arthroplasty; Anterior total hip replacement; Transient neurological symptoms; Spinal anesthesia
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine prior to THA (Active Comparator): Participants scheduled for Total Hip Arthroplasty through anterior approach with Lidocaine spinal anesthesia and completing telephone questionnaires to see how they are feeling post-operation.
  Interventions: Drug: Lidocaine
- Bupivacaine prior to THA (Active Comparator): Participants scheduled for Total Hip Arthroplasty through anterior approach with Bupivacaine spinal anesthesia and completing telephone questionnaires to see how they are feeling post-operation.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Lidocaine — Spinal anesthesia administered prior to participant's THA
  Arms: Lidocaine prior to THA
Drug: Bupivacaine — Spinal anesthesia administered prior to participant's THA
  Arms: Bupivacaine prior to THA

SUMMARY:
Spinal anesthesia is commonly used in patients undergoing total hip replacements. The purpose of this study is to compare lidocaine to bupivacaine spinal anesthesia in patients having a total hip arthroplasty (THA). The objective of this study is to compare the two spinal anesthesia treatments in regards to transient neurological symptoms (TNS).

DETAILED DESCRIPTION:
Most surgeons would agree total hip arthroplasty (THA) is one of the most successful surgical interventions. However, when it comes to the type of anesthesia to improve THA outcomes, surgeons do not agree. General anesthesia has been shown to be associated with increases in adverse events, increased operating room times and increased length of stay. Therefore, more surgeons are turning to spinal anesthesia for better pain control, decreased need for narcotics resulting in less nausea, sooner recovery of bowel function, and faster participation in physical therapy. All of these factors can lead to a sooner discharge from the hospital, which would lead to significant cost savings.

Transient neurological symptoms (TNS) are a concern of using spinal anesthesia and have been shown to occur up to 16-40% of the time with lidocaine. Symptoms of TNS have been described as pain, dysesthesia, or both that occur in the legs or buttocks and urinary retention after recovery from spinal anesthesia. Intensity of pain varies but can be quite severe. Symptoms can appear in a few hours, for up to 24 hours after surgery.

Lidocaine is the most widely used anesthetic due to its rapid onset, intense nerve blockade, and short duration of action. The risk of developing TNS after spinal anesthesia with lidocaine has been shown to be higher when compared to other anesthetics. However, it is unknown whether there are differences between patients who undergo spinal anesthesia with lidocaine versus bupivacaine in THA. This knowledge is important because it has been shown that bupivacaine spinal anesthesia is more effective than lidocaine with minimal adverse effects. A large randomized, prospective study is needed to prove the difference between the two types of anesthesia.

The primary objective of this study is to compare TNS among people who receive one of two spinal anesthesia treatments, lidocaine or bupivacaine. The study will be conducted on individuals who are indicated for THA and have agreed to have spinal anesthesia during their surgery. All patients will be randomized by a computer program and will receive either lidocaine or bupivacaine spinal anesthesia prior to their THA. In addition to TNS, other outcomes include urinary retention, hypotension, ambulation and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of symptomatic osteoarthritis in one or bilateral hips. Osteoarthritis will be defined as pain with weight-bearing at the hip articulation together with radiographic findings
* Indicated for total hip arthroplasty
* Agreement to undergo spinal anesthesia for surgery

Exclusion Criteria:

* Patient refusal to undergo spinal anesthesia
* Patients with a known history of lumbar or sacral spinal fusion.
* Patients with a known history of prostate, urological, or kidney surgery.
* Patients who need monitoring of urine output during surgery (including patients with confirmed renal disease, renal failure, chronic renal insufficiency, or an indwelling catheter at the time of surgery).
* Current infection at site of injection
* Women of child-bearing potential who are on Medicare (child-bearing potential will be determined prior to surgery per Anesthesia standard of care)
* Hypovolemia
* Indeterminate neurologic disease
* Allergy or hypersensitivity to the study medications
* Currently taking any anti-coagulation medications or coagulopathic
* Increased intracranial pressure
* Subject is unable to make his/her own decision regarding the informed consent
* Subject is unable to read/understand English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bradbury, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Orthopaedic and Spine Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lidocaine Spinal Anesthesia: Participants scheduled for total hip arthroplasty (THA) who were randomized to receive lidocaine spinal anesthesia.
- Bupivacaine Spinal Anesthesia: Participants scheduled for total hip arthroplasty (THA) who were randomized to receive bupivacaine spinal anesthesia.
Period: Overall Study
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Started | 67 | 68
Completed | 11 | 12
Not Completed | 56 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.08 (11.056) | 61.22 (10.98) | 61.13 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 66
  Male | 30 | 39 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 67 | 68 | 135

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Transient Neurological Symptoms (TNS) on Day 1 Post-Operation
Description: Following a prepared questionnaire, a study team member asked about TNS and pain that was not associated with the operation area. The count of participants reporting any type of TNS is presented here.
Time Frame: Day 1 (day of surgery) Post-Operation
Population: This analysis includes participants who completed the Neurological Symptoms Checklist. Two participants were assessed for other outcomes post-operatively on day of surgery but TNS was not evaluated. Sixteen participants were not assessed post-operatively on day of surgery for any outcomes, or their records were lost. Details about some study visits are no longer available and the exact reasons for the missing data cannot be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 48 | 50
Participants | 3 | 1

2. Primary Outcome: Post-Operative Transient Neurological Symptoms Score on Day 1 Post-Operation
Description: Following a prepared questionnaire, a study team member asked about symptoms of TNS and pain that was not associated with the operation area. Participants were asked to grade the symptoms on a verbal analogue scale from 0 to 10, with zero as no discomfort and ten as unbearable discomfort.
Time Frame: Day 1 (day of surgery) Post-Operation
Population: This analysis includes participants reporting any type of TNS following surgery, on the day of surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 3 | 1
score on a scale | 2 (1.0) | 4 (0.0)

3. Primary Outcome: Number of Participants With Transient Neurological Symptoms on Post-Operative Day 7
Description: as for outcome 1
Time Frame: Post-Operative Day 7
Population: This analysis includes participants who completed the Neurological Symptoms Checklist. One participant in the lidocaine group participated in the Post-Operative Day 7 follow-up phone call but did not complete the Neurological Symptoms Checklist. The remaining missing participants were lost to follow up, were not called for this follow-up assessment, or their records were lost. Details about some study visits are no longer available and the exact reasons for missing data cannot be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 14 | 17
Participants | 3 | 4

4. Primary Outcome: Transient Neurological Symptoms Score on Post-Operative Day 7
Description: as for outcome 2
Time Frame: Post-Operative Day 7
Population: This analysis includes participants reporting any type of TNS during the Post-Operative Day 7 follow-up assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 3 | 4
score on a scale | 2.33 (2.52) | 5.75 (4.19)

5. Primary Outcome: Number of Participants With Transient Neurological Symptoms on Post-Operative Day 14
Description: Following a prepared questionnaire, a study team member asked about symptoms of TNS and pain not associated with the operation area. The count of participants reporting any type of TNS is presented here.
Time Frame: Post-Operative Day 14
Population: This analysis includes participants who completed the Neurological Symptoms Checklist. Thirteen participants in the Bupivacaine group participated in the Post-Operative Day 14 follow-up phone call but only 12 completed the TNS assessment. The remaining missing participants were lost to follow up, were not called for the Post-Operative Day 14 assessment, or their records were lost. Details about some study visits are no longer available and the exact reasons for missing data cannot be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 11 | 12
Participants | 9 | 3

6. Primary Outcome: Transient Neurological Symptoms Score on Post-Operative Day 14
Description: as for outcome 2
Time Frame: Post-Operative Day 14
Population: This analysis includes participants reporting any type of TNS following surgery on Post-Operative Day 14.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 9 | 3
score on a scale | 2.56 (1.88) | 5.67 (3.06)

7. Secondary Outcome: Number of Participants Voiding Without Complications After Recovery From Spinal Anesthesia
Description: Urine retention after recovery from spinal anesthesia was assessed as the count of participants voiding without complications. Data were obtained through review of the inpatient records.
Time Frame: Day 1 (day of surgery) Post-Operation
Population: This analysis includes participants who had data regarding urinary voiding recorded. Details about some study visits are no longer available and the exact reasons for missing data cannot be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 48 | 50
Participants | 47 | 47

8. Secondary Outcome: Time to Ambulation After Recovery From Spinal Anesthesia
Description: Time to ambulation after recovery from spinal anesthesia is assessed in minutes. Information about time to full ambulation was obtained by asking participants or from inpatient medical charts.
Time Frame: Day 1 (day of surgery) Post-Operation
Population: This analysis includes participants who had the time when they were fully ambulatory recorded. Details about some study visits are no longer available and the exact reasons for missing data cannot be determined.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 47 | 49
minutes | 279.3 (273.0) | 242.0 (91.23)

9. Secondary Outcome: Count of Participants With Hypotension
Description: The number of participants experiencing hypotension, defined as systolic blood pressure of <90 mmHg, is presented here. Blood pressure information was obtained from reviewing the inpatient medical charts.
Time Frame: Day 1 (day of surgery) Post-Operation
Population: This analysis includes participants with post-operative blood pressure data recorded. Details about some study visits are no longer available and the exact reasons for missing data cannot be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 49 | 51
Participants | 2 | 1

10. Secondary Outcome: Number of Participants Discharged 0, 1, or 2 Days Following Surgery
Description: Hospital length of stay was obtained from inpatient charts. Length of stay was determined using the hospital admission dates and discharge dates, and was then categorized as being discharged the same day as the surgery, the day after surgery, or two days after surgery.
Time Frame: Up to Post-Operative Day 2
Population: This analysis includes participants with discharge data collected from medical records. Details about some study visits are no longer available and the exact reasons for missing data cannot be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
Number analyzed (Participants) | 49 | 51
Participants
  Day of surgery | 35 | 44
  Post-operative Day 1 | 10 | 6
  Post-operative Day 2 | 4 | 1

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the day of surgery through the 14 Days Post-Operative phone call (15 days total).
Arm/Group | Lidocaine Spinal Anesthesia | Bupivacaine Spinal Anesthesia
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68
Other Adverse Events (participants affected / at risk) | 0/67 | 0/68

LIMITATIONS AND CAVEATS:
The study was terminated due to extended suspension of the study related to personnel issues and pandemic-related issues. Missing data due to lost study records limited the number of available data points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT02818894/Prot_SAP_000.pdf